CLINICAL TRIAL: NCT05094817
Title: Feasibility of an Online, Self-administered Cognitive Screening Tool in Older Patients Undergoing Ambulatory Surgery (FOCUS)
Brief Title: Feasibility of an Online, Self-administered Cognitive Screening Tool in Older Patients Undergoing Ambulatory Surgery
Acronym: FOCUS
Status: Completed | Type: Observational
Sponsor: Women's College Hospital (Other)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-0155-E
Record Dates: First submitted 2021-07-05; First posted 2021-10-26 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Delirium in Old Age; Alzheimer Disease; Mild Cognitive Impairment; Neurocognitive Disorders
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Neurocognitive Disorders | interventions — Patient Health Questionnaire

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Access to Computer: Participants completing the BHA should be at least somewhat comfortable or very comfortable with using a computer and mouse and should use a computer at least once a week.
  Interventions: Other: Brain Health Assessment; Other: Demographics questionnaire; Other: PHQ-2; Other: AFT; Other: GAI-SF; Other: pain VAS; Other: IADL; Other: FAM CAM; Other: 4AT; Other: BHA Usability Survey; Other: Clinical Frailty Scale
- No Access to Computer: Since participants in previous studies on cognitive screening are usually more educated individuals with higher income, participants who do not have proficiency/or access to a computer will be asked to complete some questionnaires to determine any sociodemographic or baseline differences between patients who are able to complete BHA vs. those who are not able to complete BHA.
  Interventions: Other: Demographics questionnaire; Other: PHQ-2; Other: AFT; Other: GAI-SF; Other: pain VAS; Other: IADL

INTERVENTIONS:
Other: Brain Health Assessment — BHA is a free, self-administered online cognitive screening test developed in Toronto at Baycrest (www.cogniciti.com). BHA has been validated against a gold standard neuropsychological assessment for detecting amnestic MCI (aMCI) - the most common type of MCI - in community dwelling older adults. BHA has high sensitivity (.78), specificity (.78), PPV (.82), NPV (.74), and was better than MoCA for identifying aMCI. ROC curves showed an AUC of 0.75 for detecting aMCI from normal subjects. BHA measures memory and executive attention processes sensitive to subtle cognitive changes associated with normal aging and MCI. BHA can be completed from a patient's home or can be self-administered in hospital.
  Groups: Access to Computer
Other: Demographics questionnaire — To compare the sociodemographic characteristics of patients completing Cogniciti's BHA vs. those who are not able to complete the BHA.
Other: PHQ-2 — PHQ-2 is a shortened version of PHQ-9 which is originally a component of the longer Patient Health Questionnaire. The tool incorporates DSM-IV depression criteria and other leading major depressive symptoms into brief self-reported instruments. PHQ-2 inquires about the degree to which an individual experiences depression and anhedonia (inability to feel pleasure) over the past two weeks. The tool is not for final diagnosis of depression or monitoring its severity but only for the purpose of screening for the condition.The questionnaire comprises of the first two questions from PHQ-9, each item is scored 0-3. Therefore, the PHQ-2 score ranges from 0-6.
Other: AFT — AFT is a free, rapid cognitive assessment commonly used to assess semantic language ability. Language is one of the earliest functions affected by AD and naming and semantical knowledge seems to be particularly affected. The identification of language deficits may pick up signs of neurological decline preceding the appearance of clinical symptoms. Milder forms of cognitive impairment such as MCI may also show language deficits if language is one of the domains affected.
Other: GAI-SF — GAI-SF is a 5-item questionnaire derived from the original 20-item Geriatric Anxiety Inventory (GAI).In the population of community dwelling older women GAI-SF was developed in, a cut-off score of 3 yields a specificity of 87% and sensitivity of 75%. This highly accessible questionnaire is suitable for everyday use in a range of health-care settings. It has been employed amongst older adults in primary care settings, nursing homes, geriatric psychiatry patients and amongst clinical geriatric participants with co-morbid anxiety and unipolar mood disorder and their controls.
Other: pain VAS — The VAS is a unidimensional measure of pain intensity. The VAS tries to measure a continuous characteristic or attitude signifying the intensity or frequency of symptoms. The scale ranges from 0-10, with 0 = no pain to 10 = worst pain.
Other: IADL — Instrumental activities such as preparing meals or managing finances allow individuals to maintain their health while living on their own. The IADL measures the ability of older adults to manage their daily activities, as well as the impact, if any, cognitive decline would have on these activities. Scores range from 0-5 for men, and 0-8 for women, with higher sores being more independent and higher functioning.
Other: FAM CAM — FAM-CAM was derived from the CAM instrument in order to screen for delirium by interviewing family members or caregivers of the patient. They are asked specific questions about any new or sudden changes in the patient's activity, behavioural or cognitive status. FAM-CAM showed good sensitivity and specificity in the original study where caregivers of elderly patients with pre-existing cognitive impairment were interviewed.
  Groups: Access to Computer
Other: 4AT — The 4AT is a rapid tool for delirium detection that has previously been used in a surgical setting. The 4Ats test for the patient's alertness, mental state, attention, and signs of acute change. Across 17 studies, the pooled sensitivity and specificity of 4AT was 0.86 and 0.89. The 4AT will be administered after the patient has completed surgery, prior to discharge.
  Groups: Access to Computer
Other: BHA Usability Survey — The survey aims to assess system usability and acceptability based on standard questions adapted from the validated System Usability Scale. The questions evaluate satisfaction, experience with technology, and comfort level, as well as questions targeting usability concerns typically experienced by older adults, such as typeface and font size, consistent navigation, and writing style.
  Groups: Access to Computer
Other: Clinical Frailty Scale — CFS is a 9-item scale that uses clinical descriptors and pictographs and is an easily applicable tool to stratify older adults according to level of vulnerability. The CFS divides patients into 9 classes from very fit (CFS = 1) to terminally ill (CFS = 9). It is easy to use and may readily be administered in a clinical setting, an advantage over the tools previously developed. The scale helps in objective early identification of older adults with frailty in acute care units and helps to target interventions to prevent complications and to implement effective discharge planning.
  Groups: Access to Computer

SUMMARY:
Delirium is common in older adults after inpatient surgery and may be associated with cognitive decline. Advances in surgical and anesthetic techniques have led to increasing numbers of older adults undergoing surgery on an outpatient basis. However, few studies have investigated cognitive disorders of older adults before or after ambulatory surgery. Increased age and pre-existing cognitive impairment are strong risk factors for cognitive decline after surgery, yet older adults are not screened for cognitive impairment before surgery. Existing screening tools require specially trained staff for test administration and in-person testing. Virtual cognitive screening has not been evaluated in surgical patients. In this study, investigators will determine the feasibility of using Cogniciti's Brain Health Assessment (BHA) - a validated online cognitive screening tool that can be self-administered from a patient's home before surgery - to screen older adults before ambulatory surgery.

DETAILED DESCRIPTION:
Older adults (≥60 years of age) are the fastest growing age group in Canada, and by the year 2026, will constitute more than 1 of every 5 Canadians. World-wide, about 703 million people are ≥65 years of age, and this number is projected to double to 1.5 billion in 2050. Higher life expectancy and advancements in anesthetic techniques have led to more older adults with high burdens of co-morbidities to undergo ambulatory surgeries.

Approximately 40-53% of all surgeries performed are on patients >65 years of age. Neurocognitive disorders (NCD) are common in the community with 14-48% of those >age 70 years suffering mild cognitive impairment (MCI).

Impairments in cognitive ability are the most common complications in older adults undergoing major surgery. These impairments include 1) delirium (which may last up to 7 days after surgery), 2) delayed neurocognitive recovery (cognitive decline up to 30 days after surgery) 3) Neurocognitive disorder (postoperative) mild or major (30 days to 12 months after surgery). The decline in executive function, memory, and other cognitive domains may last for weeks to months after surgery. While most patients recover from cognitive impairment, a small minority of patients have persistent impairment. Older adults who are diagnosed with PND have longer hospital length of stay, are less likely to be discharged home, increased health care costs, and a higher incidence of mortality at one year after surgery.

Investigators hypothesize that it is feasible to utilize the BHA to screen for NCDs, and to assess cognitive changes in elderly patients undergoing elective ambulatory surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥65 years old)
* Undergoing elective ambulatory surgery
* Participants must be competent to provide informed consent,
* Be proficient in English (Grade 6 reading level)
* Have cognitive, visual, and physical capability necessary to complete the questionnaires and/or online assessment tool.
* Participants completing the BHA should be at least somewhat comfortable or very comfortable with using a computer and mouse and should use a computer at least once a week.

Exclusion Criteria:

* Inability to speak, read or understand English
* Previous intracranial surgery
* A previous diagnosis of major NCD e.g. dementia, and current significant uncontrolled psychiatric disorders.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients ≥65 years old from pre-operative clinics at WCH and TWH will be approached. Research personnel will identify participants that meet the inclusion criteria and informed consent will be obtained from eligible participants.
Sampling Method: Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2022-02-11 (Actual); Primary Completion 2023-07-21 (Actual); Study Completion 2023-07-21 (Actual)

PRIMARY OUTCOMES:
Participants that completed BHA/total participants | 12 months to 18 months
  To determine the feasibility (recruitment capability, rates of completion, resulting sociodemographic characteristics) of using a self-administered cognitive assessment tool (Cogniciti's BHA) in older adults undergoing elective ambulatory surgery.

SECONDARY OUTCOMES:
Usability and acceptability of Cognitici's BHA | 12 months to 18 months
  The survey aims to assess system usability and acceptability based on standard questions adapted from the validated System Usability Scale. The questions evaluate satisfaction, experience with technology, and comfort level, as well as questions targeting usability concerns typically experienced by older adults, such as typeface and font size, consistent navigation, and writing style.
Percentage of patients who successfully complete Cogniciti's BHA | 12 months to 18 months
  percentage of enrolled patients who complete all postoperative assessments
To estimate the incidence of pre-existing neurocognitive disorders (NCD) in older adults undergoing elective ambulatory surgery. | 12 months to 18 months
  Identify neurocognitive disorders among older adults undergoing ambulatory surgeries

OTHER OUTCOMES:
The sociodemographic characteristics of patients completing Cogniciti's BHA vs. those who that do not. | 12 months to 18 months
  Identify sociodemographic characteristics of patients who have been completed the BHA

CONTACTS AND LOCATIONS:
Overall Officials: Jean Wong, MD, Principal Investigator — Women's College Hospital
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Publication